CLINICAL TRIAL: NCT02819843
Title: A Phase II Randomized Trial of Intralesional Talimogene Laherparepvec (TALIMOGENE LAHERPAREPVEC) With or Without Radiotherapy for Cutaneous Melanoma, Merkel Cell Carcinoma, or Other Solid Tumors
Brief Title: A Study of T-VEC (Talimogene Laherparepvec) With or Without Radiotherapy for Melanoma, Merkel Cell Carcinoma, or Other Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-224
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-04

CONDITIONS: Melanoma; Merkel Cell Carcinoma; Other Solid Tumors
Keywords: T-VEC (Talimogene Laherparepvec); Radiotherapy; 16-224
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell | interventions — talimogene laherparepvec; Radiation Dose Hypofractionation

ARMS (2):
- Intralesional TALIMOGENE LAHERPAREPVEC with radiotherapy (Experimental): Patients will receive 3 radiotherapy treatments (one treatment every 3-5 days) during weeks 3 and 4. The first treatment will occur 6 (+/- 2) hours after the Talimogene Laherparepvec administration at week 3.Talimogene Laherparepvec will be administered at weeks 0, 3, 5, 7, 9, 11, 13 and 15. The first dose of Talimogene Laherparepvec will be 10^6 plaque forming units (PFU)/mL, followed three weeks later by a dose of 10^8 pfu/mL.
  Interventions: Drug: TALIMOGENE LAHERPAREPVEC (TVEC); Radiation: Hypofractionated Radiotherapy
- Intralesional TALIMOGENE LAHERPAREPVEC without radiotherapy (Experimental): Patients will receive Talimogene Laherparepvec alone, as described above, without radiotherapy.
  Interventions: Drug: TALIMOGENE LAHERPAREPVEC (TVEC)

INTERVENTIONS:
Drug: TALIMOGENE LAHERPAREPVEC (TVEC)
Radiation: Hypofractionated Radiotherapy
  Arms: Intralesional TALIMOGENE LAHERPAREPVEC with radiotherapy

SUMMARY:
The purpose of this phase II clinical study is to test the good and bad effects of T-VEC (talimogene laherparepvec) with or without hypofractionated radiotherapy on people with melanoma, Merkel cell carcinoma, or other solid tumors with skin metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years old
* Life expectancy > 4 months
* Histopathologically confirmed melanoma, Merkel cell carcinoma or other solid tumor malignancy
* Cutaneous subcutaneous soft tissue, or superficial lymphatic metastasis not suitable for surgical resection
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Cutaneous subcutaneous soft tissue, or superficial lymphatic metastasis that is amenable to injection and irradiation and > 10 mm in longest dimension

  ° Cutaneous metastasis in a region of previous radiation therapy is amenable to radiation therapy as part of this protocol if at least 6 months has elapsed since prior radiotherapy and the dose of radiotherapy previously administered did not exceed an equivalent dose of 60 Gy in 2 Gy equivalent fractions at the skin surface (using linear-quadratic modeling with alpha/beta=11.5)
* Metastasis that is > 10 mm in longest dimensionor exhibits radiotracer uptake consistent with metastasis on PET/CT
* Adequate coagulation function (platelet count >50 k/mcL, international normalized ratio of < 1.5)
* Resolution or stabilization of clinically significant adverse events from prior therapy
* Able to provide valid written informed consent

Exclusion Criteria:

* Active herpetic skin lesions or prior complications of HSV-1 infection (such as herpetic keratitis, herpetic encephalitis)
* Receipt of a therapeutic anticoagulant
* Receipt of live vaccine within 28 days of planned first dose of TVEC
* Receipt of another cancer therapy (targeted therapy, chemotherapy, investigational therapy, immunotherapy, radiotherapy or surgery) which is yielding an overall response (by response criteria in this study)

  ° Patients with stable or progressing disease (as determined by at least 2 consecutive assessments at 6-week interval) can continue to receive the same therapy during treatment as part of this protocol
* History of symptomatic autoimmune disease (such as lupus, scleroderma, Crohn's disease, ulcerative colitis) requiring systemic treatment (for example corticosteroids or immunosuppressants); replacement therapy (for example, thyroxine, insulin) is not considered a systemic treatment
* History of high grade (CTCAE ≥ Grade 3) immune mediated adverse event from prior cancer immunotherapy
* History of CTCAE ≥ Grade 2 immune mediated endocrinopathy from prior cancer immunotherapy
* Intermittent or chronic use of oral or intravenous antiherpetic drug (such as acyclovir)
* Active or chronic hepatitis B or C infection

  ° Previously infected, with evidence of immunity and no evidence of active hepatitis is not an exclusion criterion
* Known human immunodeficiency virus (HIV) infection
* Known leukemia or lymphoma
* Common variable immunodeficiency
* Patients requiring chronic high dose immunosuppressants including steroids (prednisone daily equivalent of ≥ 10 mg)
* Known severe congenital or acquired cellular or humoral immunodeficient or immunocompromised patients
* High likelihood of protocol non-compliance (in opinion of investigator)
* Woman of childbearing potential unwilling to use effective contraception during protocol treatment and for 3 months after last dose of Talimogene Laherparepvec
* Woman of childbearing potential that is pregnant or breast-feeding, or planning to become pregnant or breast-feed during protocol treatment and for 3 months after last dose of Talimogene Laherparepvec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intralesional TALIMOGENE LAHERPAREPVEC Without Radiotherapy: Patients will receive Talimogene Laherparepvec alone, as described above, without radiotherapy.
  TALIMOGENE LAHERPAREPVEC (TVEC)
- Intralesional TALIMOGENE LAHERPAREPVEC With Radiotherapy: Patients will receive 3 radiotherapy treatments (one treatment every 3-5 days) during weeks 3 and 4. The first treatment will occur 6 (+/- 2) hours after the Talimogene Laherparepvec administration at week 3.Talimogene Laherparepvec will be administered at weeks 0, 3, 5, 7, 9, 11, 13 and 15. The first dose of Talimogene Laherparepvec will be 10^6 plaque forming units (PFU)/mL, followed three weeks later by a dose of 10^8 pfu/mL.
  TALIMOGENE LAHERPAREPVEC (TVEC)
  Hypofractionated Radiotherapy
Period: Overall Study
Arm/Group | Intralesional TALIMOGENE LAHERPAREPVEC Without Radiotherapy | Intralesional TALIMOGENE LAHERPAREPVEC With Radiotherapy
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Disease progression before RT | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intralesional TALIMOGENE LAHERPAREPVEC Without Radiotherapy | Intralesional TALIMOGENE LAHERPAREPVEC With Radiotherapy | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Median (Full Range); unit: years] | 70 [32 to 76] | 62 [44 to 87] | 65 [32 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: Overall subject level response is defined as partial or complete (>50% or greater decrease in largest lesion) by the modified World Health Organization (mWHO) criteria, and will include measurements of tumor size by CT component of PET/CT, and clinically by digital photography.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intralesional TALIMOGENE LAHERPAREPVEC Without Radiotherapy | Intralesional TALIMOGENE LAHERPAREPVEC With Radiotherapy
Number analyzed (Participants) | 9 | 10
Participants
  Complete Response | 1 | 1
  Partial Response | 0 | 0
  Stable Disease | 2 | 5
  Progressive Disease | 6 | 4

ADVERSE EVENTS:
Time Frame: Up to 30 months
Arm/Group | Intralesional TALIMOGENE LAHERPAREPVEC Without Radiotherapy | Intralesional TALIMOGENE LAHERPAREPVEC With Radiotherapy
All-Cause Mortality (participants affected / at risk) | 8/9 | 9/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intralesional TALIMOGENE LAHERPAREPVEC Without Radiotherapy (N=9) | Intralesional TALIMOGENE LAHERPAREPVEC With Radiotherapy (N=10)
Fever (General disorders) | 5 | 3
Fatigue (General disorders) | 2 | 3
Chills (General disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 0 | 3
Pain (General disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT02819843/Prot_SAP_000.pdf